CLINICAL TRIAL: NCT04876820
Title: Study of the Impact of Pharmaceutical Interventions on the Medication Adherence of Epileptic Patients and Their Medication Knowledge
Brief Title: Impact of Pharmaceutical Interviews on the Medication Adherence of Epileptic Patients
Acronym: EPIPHARM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decesion, no inclusion since august 2022
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_84; 2021-A00578-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
Keywords: Treatment adherence; epilepsy; hospital pharmacy; clinical pharmacy; pharmacist intervention
MeSH Terms: conditions — Epilepsy; Treatment Adherence and Compliance | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist-led intervention (Experimental)
  Interventions: Other: Pharmacist intervention
- Standard of care (Sham Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Pharmacist intervention — In the intervention arm, the patient meets with the pharmacist. Pharmaceutical intervention (H1) about anti-epileptic drugs prescribed will be done: information on when to take the medication, what to do if you forget to take it or vomit, and an explanation of adverse events. The aim is to improve medication adherence and patient knowledge. A report will be sent to the community pharmacist.
  An assessment of medication adherence to antiepileptic drug by MPR at H1 3 months and 6 months (phone call to community pharmacist) will be done. The health insurance score will also be done.
  An assessment of patient knowledge by a self-made knowledge questionnaire (10 items) at H1 in pre- post interview -, 3 and 6 months (phone call to patient) will be done.
  An assessment of pharmacists' satisfaction about community hospital network by a satisfaction questionnaire will be done.
  Arms: Pharmacist-led intervention
Other: Standard of care — An assessment of medication adherence to antiepileptic drug by MPR at the inclusion then 3 months and 6 months later will be done by a phone call to the community pharmacist. An assessment of patient knowledge by a self-made knowledge questionnaire (10 items) at the inclusion then 3 and 6 months later will be done by a phone call to the patient. The health insurance score will be also done during this call.
  Arms: Standard of care

SUMMARY:
Many studies have reported a disparity in medication adherence among epileptic patients. In this population, Medication Possession Ratio (MPR) is an index of medication adherence. MPR is defined as the ratio of the number of days of treatment delivered to the number of days in the period of interest.

No-adherents patients are defined by a MPR of less than 80% , in whom an increase in seizures and the rate of hospitalization can be observed. A pharmacist-led intervention and medication information to epileptic patients could improve patient medication adherence to antiepileptic drugs, and possibly decrease the frequency of seizures, hospitalizations and the health costs generated by these hospitalizations. This intervention could also improve patient knowledge about their medications.

The aim of this study is to evaluate the effectiveness of a pharmacist-led intervention on medication adherence of epileptic patients with the MPR. Secondary objectives include the comparison of medication adherence with health insurance score, the evaluation of patients knowledges about their medications, community pharmacists' satisfaction about community hospital network, the comparison of the seizure free patient rate and the comparison of the rate of patient in whom seizure have decreased by 50%

ELIGIBILITY:
Inclusion Criteria:

* Epileptic patients seeing a neurologist in the neurophysiology clinic with a regular follow-up by the Lille University Hospital reference center
* Adult over 18 years old
* Living at home
* Socially insured patient
* In the case of cognitive problems, the presence of a reliable caregiver managing the medications

Exclusion Criteria:

* Inpatients
* Patient under curatorship, guardianship and/or institutionalized
* Dementia
* Patient who has participated in a therapeutic education program (TEP) about his epilepsy within the previous two years
* Administrative reasons: impossibility to receive informed information, impossibility to participate in the entire study, lack of coverage by the social security system, refusal to sign the consent form.
* Switching to home care by a registered nurse for treatment management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio (MPR) | at 3 months after inclusion
  Compare adherence to antiepileptic drugs between patients who received pharmacist led intervention and those who did not by Medication Possession Ratio (MPR) 3 months after inclusion

SECONDARY OUTCOMES:
Medication Possession Ratio (MPR) | at 6 months after inclusion
  Compare adherence to antiepileptic drugs between patients who received pharmacist led intervention and those who did not by Medication Possession Ratio (MPR) 6 months after inclusion
Rate of MPR >80 percent | at 3 months and 6 months
  Compare the rate of adherent patients rate (MPR > 80 percent) between the two arms at 3 and 6 months
Pharmaceutical interview measured by responses to the knowledge Questionnaire (10-point score) | at 1 hour, 3 months and 6 months
  Evaluate the development (before vs after led pharmacist intervention) and maintenance of patient knowledge of patients received pharmacist intervention and compare them to the patient knowledge who received conventional management.
Satisfaction score on a Likert scale (score 1 to 5) | at 3 months and 6 months
  Evaluate the satisfaction of community pharmacist about community hospital network by a satisfaction questionnaire in the intervention group
Assessment of health insurance score (Score 0 to 6) | at 3 months and 6 months
  Compare drug adherence via the health insurance score between the 2 arms
Rate of patients with no seizures | at 6 months
  Compare the rate of seizure free patients between the two arms
Rate of patient in whom seizure have decreased by 50 percent | at 6 months
  Compare the rate of patient in whom seizure have decreased by 50 percent between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DERAMBURE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France